CLINICAL TRIAL: NCT00968305
Title: Cytokine Production in Children With Asthma.
Brief Title: Interleukin (IL)-13 as a Marker in Pediatrics Asthma
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Byung Ho Yu, MD, Department of Immunology and Microbiology, Rush University Medical Center
Other Study IDs: L06121901
Record Dates: First submitted 2009-08-19; First posted 2009-08-28 (Estimated); Last update posted 2009-08-28 (Estimated); Status verified 2009-08

CONDITIONS: Asthma
Keywords: African American children with stable asthma; Asthma severity; Interleukin 13 from PHA stimulated PBMC; Lung function (FEV1%); Total serum IgE; Pediatrics
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Venous blood was obtained to measure total serum immunoglobulin E, radioallergosorbent test for environmental aeroallergens, and for peripheral blood mononuclear cells isolation
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children with asthma: African American children with clinically diagnosed stable asthma

SUMMARY:
Asthma is a very common childhood chronic illness and is generally more severe in African Americans. The investigators attempted to determine whether a specific immune marker is associated with lung function and asthma severity.

DETAILED DESCRIPTION:
This study examined the relationship between Interleukin (IL)-13 from phytohemagglutinin-activated polymorphonuclear blood cells and asthma severity, lung function (measured as FEV1%), and total serum IgE levels in African American children with clinically diagnosed asthma

ELIGIBILITY:
Inclusion Criteria:

* African-American race, born in the U.S.
* Age 8-15 years
* Clinical diagnosis of asthma
* Subject is able to understand and follow verbal instructions in English

Exclusion Criteria:

* Asthma exacerbation in the 4 weeks preceding the research visit
* Oral/IV steroid use in the 4 weeks preceding the research visit
* Upper or lower respiratory tract infection in the 4 weeks preceding the research visit
* Antibiotic use in the 4 weeks preceding the research visit
* Use of a short-acting bronchodilator during the 6 hours prior to spirometry (lung function testing)
* Use of a long-acting bronchodilator during the 12 hours prior to spirometry (lung function testing)

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: African-American children, ages 8 to 15 years, with clinically diagnosed asthma which had been stable for at least 4 weeks prior to enrollment in the study.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2008-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Interleukin-13 from phytohemagglutinin activated peripheral blood mononuclear cells | 7 months (from the start to completion of study. The blood was drawn at the one and only visit for each subject)

SECONDARY OUTCOMES:
Lung function measured by percent predicted forced expiratory volume in the first second (FEV1%) | 7 months (from the start to completion of study, but FEV1% was measured at the one and only visit for each subject)

CONTACTS AND LOCATIONS:
Overall Officials: Byung H Yu, MD, Principal Investigator — Rush University Medical Center, Department of Immunology and Microbiology
Locations (1):
- Rush University Medical Center; Clinic: University Consultants in Allergy and Immunology, Chicago, Illinois, United States